CLINICAL TRIAL: NCT02325037
Title: Randomized, Double-blind, Placebo-controlled, Dose-escalation Study for the Assessment of Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GLPG1837 in Healthy Subjects
Brief Title: First-in-Human Single and Multiple Dose of GLPG1837
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1837-CL-101; 2014-003853-32 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLPG1837 single dose (Experimental): Single oral dose of GLPG1837 suspension - ascending doses
  Interventions: Drug: GLPG1837 single ascending doses
- Placebo single dose (Placebo Comparator): Single oral dose of placebo suspension
  Interventions: Drug: Placebo single dose
- GLPG1837 muliple doses (Experimental): Multiple oral doses of GLPG1837 suspension - ascending doses
  Interventions: Drug: GLPG1837 multiple ascending doses
- Placebo multiple doses (Placebo Comparator): Multiple oral doses of placebo suspension
  Interventions: Drug: Placebo multiple doses

INTERVENTIONS:
Drug: GLPG1837 single ascending doses — Single dose, oral suspension
  Arms: GLPG1837 single dose
Drug: Placebo single dose — Single dose, oral suspension matching placebo
  Arms: Placebo single dose
Drug: GLPG1837 multiple ascending doses — Multiple doses, daily for 14 days, oral suspension
  Arms: GLPG1837 muliple doses
Drug: Placebo multiple doses — Multiple doses, daily for 14 days, oral suspension, matching placebo
  Arms: Placebo multiple doses

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety and tolerability after single ascending oral doses of GLPG1837 given to healthy subjects, compared to placebo. Also, the safety and tolerability of multiple ascending oral doses of GLPG1837 given to healthy subjects daily for 14 days compared to placebo, will be evaluated.

Furthermore, during the course of the study after single and multiple oral dose administrations, the amount of GLPG1837 and its metabolite present in the blood and urine (pharmacokinetics) will be characterized.

The effect of food on the pharmacokinetics of GLPG1837 and its metabolite will also be evaluated.

The potential of cytochrome P450 (CYP)3A4 induction after repeated dosing with GLPG1837 will be explored as well.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-child bearing potential between 18-50 years of age (included)
* Subjects must have a body mass index between 18-30 kg/m² (included)
* Subjects must be judged to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram and laboratory findings

Exclusion Criteria:

* A subject with a known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug
* Concurrent participation or participation within 8 weeks prior to the initial study drug administration in a drug/device or biologic investigational research study or participation within 15 weeks prior to initial study drug administration in an investigational research study with antibody administration
* A subject with active drug or alcohol abuse within 2 years prior to the initial study drug administration
* Current sexually active (and/or child wish) male; a contraception method should be used
* Pregnant or lactating women or women of childbearing potential

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1837 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of adverse events
Number of subjects with abnormal laboratory parameters | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1837 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal laboratory parameters
Number of subjects with abnormal vital signs | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1837 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal vital signs
Number of subjects with abnormal electrocardiogram | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1837 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal electrocardiograms
Number of subjects with abnormal physical examination | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1837 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal physical examination

SECONDARY OUTCOMES:
The amount of GLPG1837 and its metabolite in plasma | Between Day 1 predose and 48 hours after the (last) dose
  To characterize the amount of GLPG1837 and its metabolite in plasma over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects, fasted or fed
The amount of GLPG1837 and its metabolite in urine | Between Day 1 predose and 24 hours after the (last) dose
  To characterize the amount of GLPG1837 and its metabolite in urine over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects, fasted or fed
Ratio of 6-b-hydroxycortisol/cortisol in urine | Twelve hours before dosing on Day 1 and Day 14
  To assess the potential of CYP3A4 induction after repeated oral dosing with GLPG1837 by means of the ratio of 6-b-hydroxycortisol/cortisol in urine

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Belgium